CLINICAL TRIAL: NCT06945380
Title: mHealth App for Caregiver Instruction in Manual Therapy for Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Evaluating a Mobile Health Application Intervention for Caregiver Instruction in Manual Therapy for Chemotherapy-Induced Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Collinge and Associates, Inc. (Other); IRIS Media Inc (Other)
Responsible Party: Principal Investigator, Cindy Tofthagen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-012668; NCI-2024-04430 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-012668 (Other: Mayo Clinic Institutional Review Board); R43CA268678 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2025-04-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Massage

STUDY DESIGN:
Intervention Model Description: usual care, attention control, and intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (PNR program) (Experimental): Dyads receive access to the PNR program to perform the relaxation massage techniques consisting of site restrictions, pressure restrictions, stroke direction and stroke length at least three times in a week (TIW) over 15-20 minutes for 12 weeks.
  Interventions: Other: Internet-Based Intervention; Procedure: Massage Therapy; Other: Survey Administration
- Arm II (attention control) (Active Comparator): Dyads receive access to a comparator program to perform the relaxation massage techniques at least TIW over 15-20 minutes for 12 weeks. Dyads may optionally receive access to the PNR program following the initial 12-week study period.
  Interventions: Other: Best Practice, Comparator Program; Other: Survey Administration
- Arm III (waitlist control) (Active Comparator): Dyads receive usual care for 12 weeks. Dyads may optionally receive access to the PNR program following the initial 12-week study period.
  Interventions: Other: Best Practice, Usual Care; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice, Comparator Program — Receive access to a comparator program
  Other Names: best practice; standard of care; standard therapy
  Arms: Arm II (attention control)
Other: Best Practice, Usual Care — Receive usual care
  Other Names: best practice; standard of care; standard therapy
  Arms: Arm III (waitlist control)
Other: Internet-Based Intervention — Receive access to the PNR program
  Arms: Arm I (PNR program)
Procedure: Massage Therapy — Perform the relaxation massage techniques
  Other Names: Massage
  Arms: Arm I (PNR program)
Other: Survey Administration — Complete surveys to assess CIPN symptoms, overall well-being and quality of life, and caregiver reaction and attitudes

SUMMARY:
This clinical trial assesses the impact of a family caregiver-delivered massage technique for use in cancer survivors with chemotherapy-induced peripheral neuropathy (CIPN). CIPN is a common cancer treatment side effect that impairs quality of life and daily functioning. Aside from the relatively transient effects of chemotherapy treatment (e.g., nausea, diarrhea, vomiting, infections, fatigue, hair loss), chemotherapy can damage nervous system structures leading to long-term CIPN effects including numbness in hands or feet, "pins and needles" or sudden stabbing pains, difficulty buttoning clothing or picking up objects, loss of balance and risk of falling, difficulty driving (steering wheel, foot pedals), and increased sensitivity to heat or cold. Caregivers who lack effective strategies of supportive care are at risk of feeling helpless, overwhelmed or frustrated watching their loved one suffer. Oncology massage (OM) teaches oncology-informed modifications, adaptations and safety precautions for a cancer survivor's specific condition, treatment history and side effects. An mobile health application (app) for caregivers can teach care for CIPN using safe oncology-informed massage techniques at home. Using the Peripheral Neuropathy Relief (PNR) program in the form of relaxation may help for stress reduction, reduced CIPN symptoms, and/or an increased sense of connection with patients and their family caregiver.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age.
* Must speak and read English.
* Have internet access.
* PATIENTS: Must have received platinum and/or taxane chemotherapy for adjuvant treatment of a solid tumor.
* PATIENTS: Screens positive for moderate to severe CIPN with a 4+ on a 0-10 scale, with 0 being no numbness/tingling or pain in hands or feet and 10 being most severe imaginable.
* PATIENTS: Last chemo dose must be 6+ months in the past (symptoms persist in 30% of recipients > 6 months, this assures those with established chronicity are included, reducing likelihood of spontaneous improvement). Also, no new chemotherapy should be anticipated during the study course.
* PATIENTS: Must have internet access.
* CAREGIVERS: Members of the patient's natural social support system including spouse, intimate partner, other family member (adult child, parent, other relative), friend or other lay person designated by the patient who agrees to serve as caregiver for the activities of the project.

Exclusion Criteria:

* PATIENTS: Other potential cause of neuropathy (e.g., diabetes).
* PATIENTS: Ongoing treatment with a neuropathy-causing medication.
* PATIENTS: History of oncology massage therapy for neuropathy in the last 3 months.
* PATIENTS: Unstable lymphedema-if the patient is considered at risk of lymphedema, they can participate because level 2 pressure is deemed safe; however, if patient has had lymphedema, their condition must be declared stable by a certified lymphedema therapist (if stable, level 2 pressure is safe for this study's interventions).
* PATIENTS: Stage IV patients are excluded because many are on active medications that continue to cause or exacerbate neuropathy, and would confound results; active metastases introduce increased risks with massage; and general comfort massage for supportive care would be more indicated than targeting CIPN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in chemotherapy-induced peripheral neuropathy (CIPN) (Patient) | At baseline, 6 and 12 weeks
  Will be measured using the Chemotherapy Induced Peripheral Neuropathy Assessment Tool (CIPNAT), a 69-item questionnaire used to assess CIPN symptoms and their impact on daily activities. Scores range from 0 to 140. Higher scores indicate greater severity of neuropathy.
Change in caregiver esteem (Caregiver) | At baseline, 6 and 12 weeks
  Will be measured using the 7-item esteem subscale of the Caregiver Reaction Assessment (CRA). The 7-item caregiver esteem subscale assesses the extent to which the caregiver experiences a sense of value and satisfaction in caregiving. Items are answered on a 5-point scale where 1=strongly disagree and 5=strongly agree. Higher scores indicate more positive self-esteem.
Change in attitude toward caregiving with CIPN (Caregiver) | At baseline, 6 and 12 weeks
  Will be measured using an Attitudes toward Caregiving with CIPN questionnaire developed by the investigators. Six questions are answered on a 5-point scale where 1=not at all and 5=extremely.

SECONDARY OUTCOMES:
Change in global well-being (Patient and caregiver) | At baseline, 6 and 12 weeks
  Will be measured using the Short Form 12 version 2 (SF12v2). The SF12v2 consists of 12 questions and is used to assess health-related quality of life. Scores range from 0 to 100, with higher scores indicating better health.
Change in caregiving impact (Caregiver) | At baseline, 6 and 12 weeks
  Will be measured using the Caregiver Reaction Assessment (CRA), a 24-item scale covering five dimensions of caregiving and producing five subscale scores and a total score representing overall caregiver burden. Items are answered on a 5-point scale where 1=strongly disagree and 5=strongly agree. Higher scores generally indicate a more negative impact.
Session effects (Patient, PNR and relaxation massage groups only) | Weeks 1-12
  Will be measured using weekly reporting session symptom ratings. Within 15 minutes before and again within 15 minutes after the reporting session, patients enter Likert scaled ratings of (1) numbness in hands/fingers, (2) numbness in feet/toes, (3) tingling in hands/fingers, (4) tingling in feet/toes, (5) discomfort in hands/fingers, (6) discomfort in feet/toes. After a Reporting Session patients also rate (7) overall satisfaction with the session received. An open response question (8) invites any comments or observations about the session that they may wish to offer (to be treated as qualitative data).

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Tofthagen, PhD, RN, Principal Investigator — Mayo Clinic; William Collinge, PhD, MPH, Principal Investigator — Collinge and Associates, Inc.
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be de-identified and shared with other researchers after the findings are published, and upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 1, 2026 -indefinitely
Access Criteria: to be determined

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials